CLINICAL TRIAL: NCT02639351
Title: A Phase 1, Randomized, Observer-Blind, Dosage-Escalation Study to Evaluate the Safety and Immunogenicity of an Aluminium Hydroxide/LHD153R Adjuvanted Meningococcal C-CRM197 Conjugate Vaccine Compared to Aluminium Hydroxide Adjuvanted Meningococcal C-CRM197 Conjugate Vaccine in Healthy Adults (18-45 Years of Age).
Brief Title: Safety and Immunogenicity of an Aluminium Hydroxide/LHD153R Adjuvanted Meningococcal C-CRM197 Conjugate Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 205496; V132_01EXP (Other: Novartis); 2014-002430-31 (EudraCT Number)
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Infections, Meningococcal
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- LHD153R Formulation 1 Group (Experimental): Healthy subjects aged 18 to 45 years who received a single dose of investigational MenC-CRM vaccine adjuvanted with 12.5 ug of LHD153R.
  Interventions: Biological: Investigational MenC-CRM adjuavnted with 12.5 ug of LHD153R
- LHD153R Formulation 2 Group (Experimental): Healthy subjects aged 18 to 45 years who received a single dose of investigational MenC-CRM vaccine adjuvanted with 25 ug of LHD153R.
  Interventions: Biological: Investigational MenC-CRM adjuavnted with 25 ug of LHD153R
- LHD153R Formulation 3 Group (Experimental): Healthy subjects aged 18 to 45 years who received a single dose of investigational MenC-CRM vaccine adjuvanted with 50 ug of LHD153R.
  Interventions: Biological: Investigational MenC-CRM adjuavnted with 50 ug of LHD153R
- LHD153R Formulation 4 Group (Experimental): Healthy subjects aged 18 to 45 years who received a single dose of investigational Meningococcal C-CRM conjugate vaccine (MenC-CRM) adjuvanted with 100 ug of LHD153R.
  Interventions: Biological: Investigational MenC-CRM adjuavnted with 100 ug of LHD153R
- MenC Group (Active Comparator): Healthy subjects aged 18 to 45 years who received a single dose of MenC-CRM vaccine.
  Interventions: Biological: Meningococcal C-CRM Conjugate Vaccine (MenC-CRM)

INTERVENTIONS:
Biological: Investigational MenC-CRM adjuavnted with 12.5 ug of LHD153R — Intramuscular (IM) vaccination of 1 dose of 0.5 mL
  Arms: LHD153R Formulation 1 Group
Biological: Investigational MenC-CRM adjuavnted with 25 ug of LHD153R — IM vaccination of 1 dose of 0.5 mL
  Arms: LHD153R Formulation 2 Group
Biological: Investigational MenC-CRM adjuavnted with 50 ug of LHD153R — IM vaccination of 1 dose of 0.5 mL
  Arms: LHD153R Formulation 3 Group
Biological: Investigational MenC-CRM adjuavnted with 100 ug of LHD153R — IM vaccination of 1 dose of 0.5 mL
  Arms: LHD153R Formulation 4 Group
Biological: Meningococcal C-CRM Conjugate Vaccine (MenC-CRM) — IM vaccination of 1 dose of 0.5 mL
  Arms: MenC Group

SUMMARY:
Dosage-Escalation Study to Evaluate the Safety and Immunogenicity of an Aluminium Hydroxide/LHD153R Adjuvanted Meningococcal C-CRM197 Conjugate Vaccine in Healthy Adults (18-45 years of age).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female individuals of 18 through 45 years of age on the day of informed consent
2. Healthy volunteers with good physical and mental health status, determined on the basis of the medical history, a physical examination and the results of the screening tests as judged by the investigator
3. Individuals who have voluntarily given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry
4. Individuals who can comply with study procedures including follow-up
5. Individuals that are able to understand, read and write German language
6. Females of childbearing potential who are using an effective birth control method which they intend to use for at least 30 days after the study vaccination.

Exclusion Criteria:

1. Progressive, unstable or uncontrolled clinical conditions
2. Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study
3. Clinical conditions representing a contraindication to intramuscular vaccination and blood draws
4. Abnormal function of the immune system
5. Received immunoglobulins or any blood products within 180 days prior to informed consent
6. Received an investigational or non-registered medicinal product within 30 days prior to informed consent or intend to participate in another clinical study at any time during the conduct of this study
7. Vulnerable subjects (e.g. persons kept in detention), study personnel or an immediate family or household member of study personnel, subjects with legal incapacity or limited legal capacity
8. Any relevant deviation from the laboratory parameters at screening as judged by the investigator
9. Previously received any vaccine that included a MenC antigen
10. Previously suspected or confirmed disease caused by N. meningitides
11. Had household contact with and/or intimate exposure to an individual with culture proven MenC
12. A positive serum or urine pregnancy test prior to the study vaccine administration or are currently lactating.
13. A positive drugs-of-abuse test prior to the study vaccine administration;
14. Received any other vaccines within 30 days prior to enrolment in this study or who are planning to receive any vaccine within 30 days from the administration of study vaccines
15. Any other condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Siena E, Schiavetti F, Borgogni E, Taccone M, Faenzi E, Brazzoli M, Aprea S, Bardelli M, Volpini G, Buricchi F, Sammicheli C, Tavarini S, Bechtold V, Blohmke CJ, Cardamone D, De Intinis C, Gonzalez-Lopez A, O'Hagan DT, Nuti S, Seidl C, Didierlaurent AM, Bertholet S, D'Oro U, Medini D, Finco O. Systems analysis of human responses to an aluminium hydroxide-adsorbed TLR7 agonist (AS37) adjuvanted vaccine reveals a dose-dependent and specific activation of the interferon-mediated antiviral response. Vaccine. 2023 Jan 16;41(3):724-734. doi: 10.1016/j.vaccine.2022.12.006. Epub 2022 Dec 21. PMID 36564274
- [Derived] Gonzalez-Lopez A, Oostendorp J, Koernicke T, Fadini T, D'Oro U, Baker S, O'Hagan DT, Del Giudice G, Siena E, Finco O, Medini D. Adjuvant effect of TLR7 agonist adsorbed on aluminum hydroxide (AS37): A phase I randomized, dose escalation study of an AS37-adjuvanted meningococcal C conjugated vaccine. Clin Immunol. 2019 Dec;209:108275. doi: 10.1016/j.clim.2019.108275. Epub 2019 Oct 24. PMID 31669193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 subjects were recruited from 1 site in Germany.
Groups:
- LHD153R Formulation 1 Group: Healthy subjects aged 18 to 45 years who received a single dose of investigational Meningococcal C-CRM conjugate vaccine (MenC-CRM) adjuvanted with 12.5 ug of LHD153R.
- LHD153R Formulation 2 Group: Healthy subjects aged 18 to 45 years who received a single dose of investigational Meningococcal C-CRM conjugate vaccine (MenC-CRM) adjuvanted with 25 ug of LHD153R.
- LHD153R Formulation 3 Group: Healthy subjects aged 18 to 45 years who received a single dose of investigational Meningococcal C-CRM conjugate vaccine (MenC-CRM) adjuvanted with 50 ug of LHD153R.
- MenC Group: Healthy subjects aged 18 to 45 years who received a single dose of Meningococcal C-CRM conjugate vaccine (MenC-CRM).
Period: Overall Study
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Started | 16 | 16 | 16 | 16 | 16
Completed | 16 | 16 | 16 | 16 | 16
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group | Total
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (7.51) | 33.8 (6.89) | 34.9 (5.18) | 34.4 (6.72) | 34.4 (7.85) | 34.9 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 6 | 6 | 24
  Male | 13 | 12 | 11 | 10 | 10 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 16 | 15 | 16 | 16 | 79
  Unknown | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited Local and Systemic Adverse Events (AEs)
Description: Assessed solicited local symptoms were injection site erythema, induration, pain and swelling. Any erythema/induration/swelling = erythema/induration/swelling spreading beyond 25 millimeters (mm) of injection site. Any pain = occurrence of the symptom regardless of intensity grade. Assessed solicited systemic symptoms were arthralgia, chills, diarrhea, fatigue, fever defined as body temperature greater than or equal to (≥) 38 degrees Celsius (°C), as measured orally, headache, loss of appetite, myalgia, nausea, rash, urticaria and vomiting. Any systemic symptom = occurrence of the symptom regardless of intensity grade.
Time Frame: Within 30 minutes of vaccination (Min) at Day 1
Population: Analysis was performed on the Solicited Safety Set which included all enrolled subjects who received a study vaccination and reported solicited local and systemic symptoms.
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  Any Erythema | 0 | 0 | 0 | 0 | 0
  Any Induration | 0 | 1 | 0 | 0 | 0
  Any Pain | 1 | 0 | 1 | 1 | 0
  Any Swelling | 0 | 1 | 0 | 0 | 0
  Any Arthralgia | 0 | 0 | 0 | 0 | 0
  Any Chills | 0 | 1 | 0 | 1 | 1
  Any Diarrhea | 0 | 0 | 0 | 0 | 0
  Any Fatigue | 0 | 0 | 0 | 0 | 0
  Any Fever | 0 | 0 | 0 | 0 | 0
  Any Headache | 0 | 0 | 0 | 0 | 0
  Any Loss of Appetite | 0 | 0 | 0 | 0 | 0
  Any Myalgia | 0 | 0 | 0 | 1 | 1
  Any Nausea | 0 | 0 | 1 | 0 | 0
  Any Rash | 0 | 1 | 0 | 0 | 1
  Any Urticaria | 0 | 0 | 0 | 0 | 0
  Any Vomiting | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Any Solicited Local and Systemic AEs
Description: Assessed solicited local symptoms were injection site erythema, induration, pain and swelling. Any erythema/induration/swelling = erythema/induration/swelling spreading beyond 25 mm of injection site. Any pain = occurrence of the symptom regardless of intensity grade. Assessed solicited systemic symptoms were arthralgia, chills, diarrhea, fatigue, fever defined as body temperature ≥ 38 °C, as measured orally, headache, loss of appetite, myalgia, nausea, rash, urticaria and vomiting. Any systemic symptom = occurrence of the symptom regardless of intensity grade. Other solicited data included: Analgesic/Antipyretics Use.
Time Frame: From Day 1 to Day 4 (excluding 30 minutes immediately after vaccination)
Population: Analysis was performed on the Solicited Safety Set which included all enrolled subjects who received a study vaccination and reported local and systemic symptoms
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  Any Erythema | 0 | 0 | 0 | 0 | 0
  Any Induration | 0 | 1 | 0 | 0 | 0
  Any Pain | 16 | 16 | 16 | 16 | 16
  Any Swelling | 1 | 2 | 0 | 0 | 0
  Any Arthralgia | 0 | 1 | 0 | 4 | 0
  Any Chills | 0 | 1 | 1 | 2 | 0
  Any Diarrhea | 0 | 0 | 1 | 2 | 0
  Any Fatigue | 3 | 2 | 3 | 5 | 3
  Any Fever | 0 | 1 | 0 | 1 | 0
  Any Headache | 3 | 6 | 3 | 5 | 8
  Any Loss of Appetite | 0 | 1 | 2 | 1 | 0
  Any Myalgia | 0 | 1 | 0 | 3 | 2
  Any Nausea | 0 | 2 | 1 | 1 | 0
  Any Rash | 0 | 0 | 0 | 0 | 0
  Any Urticaria | 1 | 0 | 0 | 1 | 0
  Any Vomiting | 0 | 0 | 1 | 1 | 0
  Analgesic/Antipyretics Use | 1 | 2 | 1 | 2 | 0

3. Primary Outcome: Number of Subjects With Any Solicited Local and Systemic AEs
Description: Assessed solicited local symptoms were injection site erythema, induration, pain and swelling. Any erythema/induration/swelling = erythema/induration/swelling spreading beyond 25 mm of injection site. Any pain = occurrence of the symptom regardless of intensity grade. Assessed solicited systemic symptoms were arthralgia, chills, diarrhea, fatigue, fever defined as body temperature ≥ 38 °C, as measured orally, headache, loss of appetite, myalgia, nausea, rash, urticaria and vomiting. Any systemic symptom = occurrence of the symptom regardless of intensity grade.
Time Frame: From Day 5 to Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  Any Erythema | 0 | 0 | 0 | 0 | 0
  Any Induration | 0 | 0 | 0 | 0 | 0
  Any Pain | 16 | 16 | 16 | 16 | 16
  Any Swelling | 0 | 0 | 0 | 0 | 0
  Any Arthralgia | 0 | 0 | 0 | 0 | 0
  Any Chills | 0 | 0 | 0 | 2 | 0
  Any Diarrhea | 0 | 0 | 0 | 1 | 0
  Any Fatigue | 1 | 1 | 0 | 4 | 0
  Any Fever | 0 | 0 | 0 | 1 | 0
  Any Headache | 4 | 3 | 2 | 5 | 2
  Any Loss of Appetite | 0 | 0 | 0 | 3 | 0
  Any Myalgia | 0 | 0 | 0 | 2 | 0
  Any Nausea | 0 | 0 | 0 | 2 | 0
  Any Rash | 0 | 0 | 0 | 0 | 0
  Any Urticaria | 0 | 0 | 0 | 0 | 0
  Any Vomiting | 0 | 0 | 0 | 1 | 0
  Analgesic/Antipyretics Use | 2 | 2 | 0 | 2 | 1

4. Primary Outcome: Number of Subjects With Any Solicited Local and Systemic AEs
Description: as for outcome 2
Time Frame: From Day 8 to Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  Any Erythema | 0 | 0 | 0 | 0 | 0
  Any Induration | 0 | 0 | 0 | 0 | 0
  Any Pain | 16 | 16 | 16 | 16 | 16
  Any Swelling | 0 | 0 | 0 | 0 | 0
  Any Arthralgia | 1 | 0 | 0 | 0 | 0
  Any Chills | 0 | 0 | 0 | 0 | 0
  Any Diarrhea | 1 | 0 | 0 | 0 | 0
  Any Fatigue | 2 | 1 | 0 | 2 | 0
  Any Fever | 1 | 0 | 0 | 1 | 0
  Any Headache | 4 | 1 | 1 | 2 | 4
  Any Loss of Appetite | 1 | 0 | 0 | 2 | 0
  Any Myalgia | 1 | 0 | 0 | 1 | 0
  Any Nausea | 1 | 0 | 0 | 1 | 1
  Any Rash | 0 | 0 | 0 | 0 | 0
  Any Urticaria | 0 | 0 | 0 | 0 | 0
  Any Vomiting | 0 | 0 | 0 | 0 | 0
  Analgesic/Antipyretics Use | 1 | 2 | 0 | 3 | 1

5. Primary Outcome: Number of Subjects With Any Solicited Local and Systemic AEs
Description: as for outcome 2
Time Frame: From Day 1 to Day 8 (excluding 30 minutes immediately after vaccination)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  Any Erythema | 0 | 0 | 0 | 0 | 0
  Any Induration | 0 | 1 | 0 | 0 | 0
  Any Pain | 16 | 16 | 16 | 16 | 16
  Any Swelling | 1 | 2 | 0 | 0 | 0
  Any Arthralgia | 0 | 1 | 0 | 4 | 0
  Any Chills | 0 | 1 | 1 | 4 | 0
  Any Diarrhea | 0 | 0 | 1 | 3 | 0
  Any Fatigue | 3 | 2 | 3 | 6 | 3
  Any Fever | 0 | 1 | 0 | 1 | 0
  Any Headache | 5 | 7 | 5 | 5 | 10
  Any Loss of Appetite | 0 | 1 | 2 | 3 | 0
  Any Myalgia | 0 | 1 | 0 | 5 | 2
  Any Nausea | 0 | 2 | 1 | 2 | 0
  Any Rash | 0 | 0 | 0 | 0 | 0
  Any Urticaria | 1 | 0 | 0 | 1 | 0
  Any Vomiting | 0 | 0 | 1 | 2 | 0
  Analgesic/Antipyretics Use | 2 | 3 | 1 | 3 | 1

6. Primary Outcome: Number of Subjects With Any Solicited Local and Systemic AEs
Description: as for outcome 2
Time Frame: From Day 1 to Day 14 (excluding 30 minutes immediately after any vaccination)
Population: Analysis was performed on the Solicited Safety Set which included all enrolled subjects who received a study vaccination and provided post-vaccination solicited local and systemic symptoms data
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  Any Erythema | 0 | 0 | 0 | 0 | 0
  Any Induration | 0 | 1 | 0 | 0 | 0
  Any Pain | 16 | 16 | 16 | 16 | 16
  Any Swelling | 1 | 2 | 0 | 0 | 0
  Any Arthralgia | 1 | 1 | 0 | 4 | 0
  Any Chills | 0 | 1 | 1 | 4 | 0
  Any Diarrhea | 1 | 0 | 1 | 3 | 0
  Any Fatigue | 3 | 2 | 3 | 6 | 3
  Any Fever | 1 | 1 | 0 | 1 | 0
  Any Headache | 6 | 7 | 5 | 5 | 10
  Any Loss of Appetite | 1 | 1 | 2 | 4 | 0
  Any Myalgia | 1 | 1 | 0 | 5 | 2
  Any Nausea | 1 | 2 | 1 | 3 | 1
  Any Rash | 0 | 0 | 0 | 0 | 0
  Any Urticaria | 1 | 0 | 0 | 1 | 0
  Any Vomiting | 0 | 0 | 1 | 2 | 0
  Analgesic/Antipyretics Use | 2 | 3 | 1 | 4 | 1

7. Primary Outcome: Number of Subjects With Any Unsolicited AEs
Description: An adverse event (AE) is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product at any dose that does not necessarily have to have a causal relationship with this treatment. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product. This definition includes intercurrent illnesses or injuries and exacerbation of pre-existing conditions. Unsolicited adverse event were defined as symptoms that were not solicited using a Subject Diary and that were spontaneously communicated by a subject who has signed the informed consent. Unsolicited AEs were collected through the Day 29 visit and the analysis was performed for Day 1-29 time frame, instead of Day 1-14 as required by protocol.
Time Frame: From Day 1 to Day 29
Population: Analysis was performed on the Unsolicited Safety Set which included all enrolled subjects who received a study vaccination and provided post-vaccination unsolicited adverse event data.
Measure: Count of Participants; unit: Participants
Groups:
- MenC Group: Healthy subjects aged 18 to 45 years who received a single dose of MenC-CRM.
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants | 4 | 2 | 1 | 4 | 4

8. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs), Medically Attended AEs (MAAEs), AEs Leading to Study Withdrawal, New Onset of Chronic Disease (NOCDs) and Adverse Events of Special Interest (AESIs).
Description: SAEs are untoward medical occurrences that at any dose resulted in death,was life-threatening,required/prolonged hospitalization,persistent/significant disability/incapacity,congenital anomaly/in important & significant medical event that could jeopardize the subject/could required intervention to prevent one of the other outcomes mentioned above.MAAEs are AEs that lead to a visit to a healthcare provider.NOCDs are adverse events that represent new diagnosis of a chronic medical condition that was not present/suspected in a subject prior to study enrolment.AESIs were defined according to MedDRA preferred terms.Certain AESIs are monitored after administration of immunostimulatory agents.These are pre-defined & include AEs in the SOCs of Gastrointestinal disorders,Liver disorders,Metabolic diseases,Musculo-skeletal disorders,Neuroinflammatory disorders,Skin disorders,Vasculitides & others.
Time Frame: From Day 1 to Day 366
Population: Analysis was performed on the Unsolicited Safety Set which included all enrolled subjects who received a study vaccination and had post-vaccination unsolicited adverse events data. Data for this endpoint was analyzed from Day 1 to study termination (Day 366). Data from day of signed informed consent till Day 1(as per protocol) were not collected.
Measure: Count of Participants; unit: Participants
Groups:
- MenC Group: Healthy subjects aged 18 to 45 years who received a single dose of MenC-CRM vaccine .
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  Any SAEs | 0 | 0 | 0 | 0 | 1
  Any MAAEs | 6 | 9 | 5 | 8 | 8
  Any AEs leading to withdrawal | 0 | 0 | 0 | 0 | 0
  Any NOCDs | 0 | 0 | 0 | 0 | 0
  Any AESIs | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Subjects With Any SAEs, MAAEs, AEs Leading to Study Withdrawal, NOCDs and AESIs.
Description: SAEs were defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required or prolonged hospitalization, persistent or significant disability/incapacity, congenital anomaly or in an important and significant medical event that could jeopardize the subject or could requiered intervention to prevent one of the other outcomes mentioned above. MAAEs were defined as an AE that lead to a visit to a healthcare provider. NOCDs were defined as AEs leading to study or vaccine withdrawal. AESIs were defined according to MedDRA preferred terms.Certain AEs of special interest (AESIs) are monitored after the administration of immunostimulatory agents. These are pre-defined and include AEs in the SOCs of Gastrointestinal disorders, Liver disorders, Metabolic diseases, Musculo-skeletal disorders, Neuroinflammatory disorders, Skin disorders, Vasculitides and others
Time Frame: From Day 1 to Day 29
Population: Analysis was performed on the Unsolicited Safety Set which included all enrolled subjects who received a study vaccination and had post-vaccination unsolicited adverse event data.
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  Any SAEs | 0 | 0 | 0 | 0 | 0
  Any MAAEs | 2 | 0 | 0 | 3 | 0
  Any AEs leading to withdrawal | 0 | 0 | 0 | 0 | 0
  Any NOCDs | 0 | 0 | 0 | 0 | 0
  Any AESIs | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Subjects With Any SAEs, MAAEs, AEs Leading to Study Withdrawal, NOCDs and AESIs.
Description: SAEs were defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required or prolonged hospitalization, persistent or significant disability/incapacity, congenital anomaly or in an important and significant medical event that could jeopardize the subject or could requiered intervention to prevent one of the other outcomes mentioned above. MAAEs were defined as an AE that lead to a visit to a healthcare provider. NOCDs were defined as AEs leading to study or vaccine withdrawal. AESIs were defined according to MedDRA preferred terms.Certain AEs of special interest (AESIs) are monitored after the administration of immunostimulatory agents. These are pre-defined and include AEs in the SOCs of Gastroin-testinal disorders, Liver disorders, Metabolic diseases, Musculo-skeletal disorders, Neuroinflammatory disorders, Skin disorders, Vasculitides and others
Time Frame: From Day 29 up to study end (Day 366)
Population: Analysis was performed on the Unsolicited Safety Set which included all enrolled subjects who received a study vaccination and had post-vaccination unsolicited adverse events data.
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  Any SAEs | 0 | 0 | 0 | 0 | 1
  Any MAAEs | 5 | 9 | 5 | 5 | 8
  Any AEs leading to withdrawal | 0 | 0 | 0 | 0 | 0
  Any NOCDs | 0 | 0 | 0 | 0 | 0
  Any AESIs | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Absolute Values for Clinical Serum Chemistry Parameters- Sodium (Na), Potassium (K), Chlorine (Cl), Blood Urea Nitrogen (BUN) and Bicarbonate.
Description: Analysis was performed on blood samples collected at Day 1 (pre-dose) for the following parameters: Na, K, Cl, BUN and bicarbonate in millimoles per liter (mmol/L).
Time Frame: At Day 1 (pre-dose)
Population: Analysis was performed on the Safety Set which included all enrolled subjects who received a study vaccination and had available safety laboratory data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
mmol/L
  Na | 138.07 (1.226) | 136.77 (1.514) | 136.73 (1.891) | 138.29 (1.875) | 137.06 (1.821)
  K | 4.253 (0.325) | 4.176 (0.162) | 4.185 (0.346) | 3.962 (0.178) | 4.253 (0.253)
  Cl | 104.25 (1.382) | 103.94 (2.057) | 103.91 (1.973) | 104.99 (2.168) | 104.03 (2.120)
  BUN | 4.545 (1.085) | 5.048 (1.422) | 5.247 (1.039) | 4.616 (0.930) | 4.606 (1.327)
  Bicarbonate | 25.42 (1.638) | 25.75 (1.293) | 27.09 (2.180) | 26.64 (1.944) | 25.98 (1.749)

12. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 1 (post-dose) for the following parameters: Na, K, Cl, BUN and bicarbonate in mmol/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: Analysis was performed on the Overall Safety Set which included all enrolled subjects who received a study vaccination and had available safety laboratory data
Measure: Mean (Standard Deviation); unit: Difference of mmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of mmol/L
  Na | -0.34 (1.051) | 0.45 (1.693) | -0.33 (2.097) | -0.86 (1.744) | -0.09 (2.020)
  K | 0.002 (0.361) | 0.043 (0.205) | 0.100 (0.310) | 0.028 (0.208) | 0.178 (0.254)
  Cl | -0.55 (1.526) | -0.32 (2.005) | -0.74 (2.080) | -1.06 (2.828) | -0.10 (2.122)
  BUN | -0.209 (0.944) | -0.911 (0.838) | -0.949 (0.940) | -0.556 (0.493) | -0.433 (0.616)
  Bicarbonate | 0.09 (1.080) | 0.51 (1.381) | 0.88 (1.690) | 0.41 (1.413) | 0.66 (1.733)

13. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 8 for the following parameters: Na, K, Cl, BUN and bicarbonate in mmol/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 8 results.
Time Frame: At Day 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of mmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of mmol/L
  Na | -0.39 (2.129) | 0.08 (2.066) | 0.68 (1.951) | -0.61 (2.305) | 0.11 (1.676)
  K | -0.030 (0.302) | 0.233 (0.274) | 0.143 (0.322) | 0.128 (0.137) | 0.071 (0.208)
  Cl | -1.37 (1.740) | -0.28 (2.467) | 0.27 (2.265) | -1.73 (4.390) | -1.30 (2.642)
  BUN | 0.125 (1.177) | -0.507 (0.758) | -0.128 (1.236) | 0.144 (1.144) | 0.003 (0.909)
  Bicarbonate | 1.20 (1.747) | 1.00 (1.485) | 0.14 (1.614) | 0.82 (1.633) | 0.41 (2.117)

14. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 29 for the following parameters: Na, K, Cl, BUN and bicarbonate in mmol/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 29 results.
Time Frame: At Day 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of mmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of mmol/L
  Na | 0.06 (1.834) | 1.11 (1.993) | 1.66 (2.317) | 0.09 (1.880) | 0.76 (1.926)
  K | -0.008 (0.426) | 0.290 (0.369) | 0.147 (0.377) | 0.204 (0.255) | 0.109 (0.299)
  Cl | -1.02 (2.144) | -0.34 (2.379) | -1.38 (1.438) | -1.21 (1.870) | -1.03 (1.862)
  BUN | 0.500 (1.199) | -0.103 (1.180) | 0.021 (1.214) | 0.476 (0.784) | 0.216 (1.023)
  Bicarbonate | 0.64 (1.672) | 2.66 (1.787) | 2.01 (2.158) | 0.52 (2.030) | 1.27 (2.340)

15. Primary Outcome: Absolute Values for Clinical Serum Chemistry Parameters-Creatinine
Description: Analysis was performed on blood samples collected at Day 1 (pre-dose) for the following parameter: Creatinine (CREA) in micro mole per liter (μmol/L)
Time Frame: At Day 1 (pre-dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
μmol/L | 77.52 (12.517) | 72.25 (12.336) | 80.43 (10.086) | 74.43 (13.459) | 74.29 (9.206)

16. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 1 (post-dose) for the following parameter: CREA in μmol/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of μmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of μmol/L | 0.64 (3.393) | 2.59 (2.622) | 0.21 (7.479) | -0.50 (4.654) | 1.41 (4.663)

17. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 8 for the following parameter: CREA in μmol/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 8 results.
Time Frame: At Day 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of μmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of μmol/L | 3.61 (5.109) | 3.48 (5.377) | 2.49 (4.936) | 2.03 (5.052) | 2.40 (3.440)

18. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 29 for the following parameter: CREA in μmol/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 29 results.
Time Frame: At Day 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of μmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of μmol/L | 4.51 (4.557) | 5.68 (5.878) | 3.09 (6.345) | 1.72 (4.906) | 3.24 (6.355)

19. Primary Outcome: Absolute Values for Clinical Serum Chemistry Parameters- Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)
Description: Analysis was performed on blood samples collected at Day 1 (pre-dose) for the following parameters: ALT and AST in International Units per liter (IU/L).
Time Frame: At Day 1 (pre-dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
IU/L
  ALT | 26.75 (11.906) | 20.17 (9.875) | 21.14 (7.920) | 22.97 (8.747) | 25.86 (12.631)
  AST | 23.30 (5.880) | 25.01 (5.058) | 24.11 (4.809) | 23.08 (6.592) | 24.84 (5.771)

20. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 1 (post-dose) for the following parameters: ALT and AST in IU/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of IU/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of IU/L
  ALT | -2.29 (3.044) | -1.28 (1.563) | -1.40 (2.892) | -1.19 (3.969) | 0.23 (2.569)
  AST | -2.41 (2.461) | -2.82 (2.451) | -3.07 (3.280) | -1.98 (3.391) | -1.44 (2.590)

21. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 8 for the following parameters: ALT and AST in IU/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 8 results.
Time Frame: At Day 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of IU/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of IU/L
  ALT | 0.70 (5.806) | 2.08 (5.027) | 0.47 (4.580) | 1.03 (6.764) | 1.88 (4.150)
  AST | 2.58 (4.930) | 2.47 (13.382) | 0.21 (6.431) | 0.43 (6.743) | 0.00 (4.103)

22. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 29 for the following parameters: ALT and AST in IU/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 29 results.
Time Frame: At Day 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of IU/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of IU/L
  ALT | -2.15 (9.553) | 2.36 (6.040) | 5.99 (10.114) | 0.91 (7.192) | 3.78 (8.382)
  AST | 0.56 (6.031) | 1.88 (16.060) | 2.24 (5.948) | -0.74 (6.674) | 2.61 (6.823)

23. Primary Outcome: Absolute Values for Clinical Serum Chemistry Parameters- C-reactive Protein (CRP)
Description: Analysis was performed on blood samples collected at Day 1 (pre-dose) for the following parameter: CRP in milligram per liter (mg/L).
Time Frame: At Day 1 (pre-dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 15 | 16 | 16
mg/L | 1.382 (3.353) | 0.928 (0.663) | 1.049 (1.003) | 2.337 (3.718) | 1.243 (1.340)

24. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 1 (post-dose) for the following parameters: CRP in mg/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of mg/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 15 | 16 | 16
Difference of mg/L | -0.148 (1.334) | 0.888 (2.177) | 0.439 (1.015) | 1.646 (4.231) | 0.239 (0.777)

25. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 8 for the following parameter: CRP in mg/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 8 results.
Time Frame: At Day 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of mg/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 15 | 16 | 16
Difference of mg/L | -0.393 (3.260) | 0.339 (0.878) | -0.057 (0.830) | 7.736 (30.996) | 0.153 (0.934)

26. Primary Outcome: Changes in Clinical Serum Chemistry Parameters
Description: Analysis was performed on blood samples collected at Day 29 for the following parameter: CRP in mg/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 29 results.
Time Frame: At Day 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Difference of mg/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 15 | 16 | 16
Difference of mg/L | -0.202 (3.195) | 0.348 (0.849) | 0.200 (0.535) | 1.075 (8.004) | -0.058 (0.948)

27. Primary Outcome: Absolute Values for Hematology Parameters- Basophils, Eosniophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Plateletes.
Description: Analysis was performed on blood samples collected at Day 1 (pre-dose) for the following parameters: basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets in 10^9 cells per liter (10^9/L)
Time Frame: At Day 1 (pre-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
10^9/L
  Basophil | 0.033 (0.015) | 0.034 (0.020) | 0.033 (0.014) | 0.030 (0.014) | 0.029 (0.012)
  Eosinophils | 0.128 (0.065) | 0.183 (0.127) | 0.184 (0.114) | 0.150 (0.105) | 0.234 (0.136)
  Leukocytes | 6.150 (2.116) | 5.278 (1.170) | 6.085 (1.720) | 6.031 (1.560) | 6.383 (1.347)
  Lymphocytes | 1.653 (0.453) | 1.764 (0.425) | 0.425 (0.562) | 1.751 (0.332) | 1.868 (0.413)
  Monocytes | 0.413 (0.110) | 0.365 (0.108) | 0.428 (0.114) | 0.398 (0.090) | 0.451 (0.115)
  Neutrophils | 3.811 (1.865) | 2.833 (0.712) | 3.502 (1.157) | 3.618 (1.372) | 3.692 (1.095)
  Platelets | 203.9 (37.90) | 208.3 (38.82) | 239.9 (60.28) | 197.8 (45.04) | 224.0 (50.46)

28. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 1 (post-dose) for the following parameters: basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets in 10^9/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of 10^9/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of 10^9/L
  Basophils | 0.000 (0.014) | 0.000 (0.009) | -0.003 (0.009) | 0.004 (0.014) | 0.001 (0.011)
  Eosinophils | 0.015 (0.045) | -0.018 (0.057) | -0.009 (0.041) | -0.016 (0.050) | 0.016 (0.052)
  Leukocytes | 0.853 (1.442) | 0.923 (1.291) | 0.584 (1.048) | 0.294 (1.531) | 0.621 (0.968)
  Lymphocytes | 0.077 (0.314) | -0.147 (0.533) | -0.302 (0.358) | -0.197 (0.397) | 0.000 (0.246)
  Monocytes | 0.075 (0.068) | 0.053 (0.102) | 0.049 (0.084) | 0.051 (0.102) | 0.040 (0.078)
  Neutrophils | 0.686 (1.436) | 1.044 (0.945) | 0.863 (0.851) | 0.451 (1.182) | 0.558 (0.873)
  Platelets | -2.5 (11.08) | -0.6 (15.19) | -0.1 (12.75) | -2.3 (9.74) | -0.8 (14.20)

29. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 8 for the following parameters: basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets in 10^9/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 8 results.
Time Frame: At Day 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of 10^9/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of 10^9/L
  Basophils | -0.001 (0.016) | 0.004 (0.010) | -0.002 (0.014) | 0.006 (0.013) | 0.006 (0.016)
  Eosinophils | 0.044 (0.048) | -0.006 (0.059) | -0.013 (0.058) | 0.025 (0.064) | 0.033 (0.074)
  Leukocytes | 0.123 (1.624) | 0.086 (0.968) | -0.417 (1.161) | -0.451 (1.245) | 0.074 (0.978)
  Lymphocytes | 0.333 (0.416) | 0.029 (0.404) | -0.007 (0.476) | 0.115 (0.349) | 0.025 (0.339)
  Monocytes | 0.004 (0.086) | -0.001 (0.069) | -0.053 (0.087) | -0.016 (0.097) | 0.027 (0.081)
  Neutrophils | -0.256 (1.567) | 0.048 (0.640) | -0.342 (0.854) | -0.603 (1.184) | -0.031 (1.015)
  Platelets | 28.2 (27.77) | 25.3 (16.19) | 13.1 (28.34) | 17.9 (16.39) | 22.4 (22.90)

30. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 29 for the following parameters: basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets in 10^9/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 29 results.
Time Frame: At Day 29
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of 10^9/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of 10^9/L
  Basophils | 0.007 (0.012) | 0.002 (0.010) | 0.003 (0.011) | 0.006 (0.012) | 0.004 (0.013)
  Eosinophils | 0.039 (0.063) | -0.014 (0.107) | 0.027 (0.078) | 0.020 (0.052) | 0.018 (0.063)
  Leukocytes | 0.136 (1.637) | 0.328 (0.781) | -0.023 (1.442) | -0.212 (1.264) | -0.086 (1.161)
  Lymphocytes | 0.294 (0.506) | 0.038 (0.476) | -0.041 (0.451) | 0.122 (0.429) | 0.105 (0.268)
  Monocytes | 0.079 (0.109) | 0.025 (0.090) | -0.002 (0.098) | -0.028 (0.099) | 0.019 (0.092)
  Neutrophiles | -0.276 (1.431) | 0.277 (0.611) | -0.016 (0.970) | -0.355 (1.228) | -0.234 (1.091)
  Platelets | 19.6 (33.37) | 24.5 (15.30) | 6.6 (15.68) | 10.1 (16.55) | 11.1 (22.47)

31. Primary Outcome: Absolute Values for Hematology Parameters- Red Blood Cells (RBC)
Description: Analysis was performed on blood samples collected at Day 1 (pre-dose) for the following parameter: RBC in 10^12 cells per liter (10^12/L).
Time Frame: At Day 1 (pre-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^12/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
10^12/L | 4.777 (0.358) | 4.598 (0.377) | 4.724 (0.492) | 4.676 (0.362) | 4.773 (0.315)

32. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 1 (post-dose) for the following parameter: RBC in 10^12/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of 10^12/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of 10^12/L | 0.024 (0.146) | 0.064 (0.198) | 0.139 (0.167) | 0.019 (0.205) | 0.069 (0.174)

33. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 8 for the following parameter: RBC in 10^12/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 8 results.
Time Frame: At Day 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of 10^12/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of 10^12/L | 0.058 (0.171) | 0.102 (0.256) | 0.014 (0.216) | 0.008 (0.144) | 0.061 (0.211)

34. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 29 for the following parameter: RBC in 10^12/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 29 results.
Time Frame: At Day 29
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of 10^12/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of 10^12/L | 0.094 (0.239) | 0.209 (0.187) | 0.197 (0.208) | -0.001 (0.200) | 0.052 (0.199)

35. Primary Outcome: Absolute Values for Hematology Parameters- Hematocrit
Description: Analysis was performed on blood samples collected at Day 1 (pre-dose) for the following parameter: hematocrit in liter per liter (L/L).
Time Frame: At Day 1 (pre-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
L/L | 0.428 (0.026) | 0.415 (0.032) | 0.409 (0.029) | 0.411 (0.033) | 0.424 (0.029)

36. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 1 (post-dose) for the following parameter: hematocrit in L/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of L/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of L/L | 0.002 (0.013) | 0.002 (0.017) | 0.013 (0.017) | -0.001 (0.019) | 0.006 (0.018)

37. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 8 for the following parameter: hematocrit in L/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 8 results.
Time Frame: At Day 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of L/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of L/L | 0.006 (0.015) | 0.010 (0.022) | 0.002 (0.018) | -0.001 (0.011) | 0.005 (0.019)

38. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 29 for the following parameter: hematocrit in L/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 29 results.
Time Frame: At Day 29
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of L/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of L/L | 0.008 (0.023) | 0.021 (0.017) | 0.021 (0.019) | 0.001 (0.016) | 0.007 (0.016)

39. Primary Outcome: Absolute Values for Hematology Parameters- Hemoglobin (HGB)
Description: Analysis was performed on blood samples collected at Day 1 (pre-dose) for the following parameter: HGB in gram per liter (g/L).
Time Frame: At Day 1 (pre-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
g/L | 144.3 (8.50) | 139.2 (11.35) | 137.1 (11.47) | 139.3 (13.15) | 143.5 (10.85)

40. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 1 (post-dose) for the following parameter: HGB in g/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of g/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of g/L | 1.6 (3.67) | 2.3 (5.43) | 4.6 (4.18) | 0.6 (5.70) | 2.3 (4.51)

41. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 8 for the following parameter: HGB in g/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 8 results.
Time Frame: At Day 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of g/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of g/L | 1.5 (5.07) | 3.8 (7.04) | 1.4 (6.15) | 2.8 (4.02) | 2.8 (4.99)

42. Primary Outcome: Changes in Hematology Parameters
Description: Analysis was performed on blood samples collected at Day 29 for the following parameter: HGB in g/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 29 results.
Time Frame: At Day 29
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of g/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of g/L | 1.2 (5.33) | 5.4 (5.55) | 5.4 (5.25) | 3.1 (4.22) | 1.6 (5.03)

43. Primary Outcome: Absolute Values for Urinalysis Parameters- Urine Erythrocytes (Urine RBC)
Description: Analysis was performed on urine samples collected at Day 1 (pre-dose) for the following parameter: Urine RBC in microliters (μL).
Time Frame: At Day 1 (pre-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: μL
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
μL | 2.8 (6.82) | 1.3 (3.42) | 7.2 (13.41) | 20.0 (20.0) | 6.9 (17.02)

44. Primary Outcome: Changes in Urinalysis Parameters
Description: Analysis was performed on urine samples collected at Day 1 (post-dose) for the following parameter: Urine RBC in μL. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of μL
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of μL | -1.6 (4.37) | 4.1 (10.52) | 5.9 (26.28) | -14.7 (58.15) | -5.6 (13.65)

45. Primary Outcome: Changes in Urinalysis Parameters
Description: Analysis was performed on urine samples collected at Day 8 for the following parameter: Urine RBC in μL. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 8 results.
Time Frame: At Day 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of μL
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of μL | -0.6 (2.50) | 1.6 (5.69) | -5.0 (12.65) | -8.4 (69.92) | 0.0 (0.00)

46. Primary Outcome: Changes in Urinalysis Parameters
Description: Analysis was performed on urine samples collected at Day 29 for the following parameter: Urine RBC in μL. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 29 results.
Time Frame: At Day 29
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of μL
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of μL | -1.3 (3.42) | 3.1 (8.14) | -1.3 (17.46) | -14.7 (64.92) | -3.8 (12.58)

47. Primary Outcome: Absolute Values for Urinalysis Parameters- Urine Glucose
Description: The absolute value for urinalysis was assessed for the following parameter: urine glucose in mmol/L.
Time Frame: At Day 1 (pre-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
mmol/L | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

48. Primary Outcome: Changes in Urinalysis Parameters
Description: Analysis was performed on urine samples collected at Day 1 (post-dose) for the following parameter: urine glucose in mmol/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: Analysis was performed on the Overall Safety Set which included all enrolled subjects who received a study vaccination and had either post-vaccination AE or reactogenicity records.
Measure: Mean (Standard Deviation); unit: Difference of mmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of mmol/L | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

49. Primary Outcome: Changes in Urinalysis Parameters
Description: Analysis was performed on urine samples collected at Day 8 (post-dose) for the following parameter: urine glucose in mmol/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 8 (post-dose) results.
Time Frame: At Day 8
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Difference of mmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of mmol/L | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

50. Primary Outcome: Changes in Urinalysis Parameters
Description: Analysis was performed on urine samples collected at Day 29 (post-dose) for the following parameter: Urine glucose in mmol/L. The change was calculated as difference between the Day 1 (pre-dose) results and the Day 29 (post-dose) results.
Time Frame: At Day 29
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Difference of mmol/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of mmol/L | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

51. Primary Outcome: Absolute Values for Urinalysis Parameters- Urine Protein
Description: The absolute value for urinalysis was assessed for the following parameter: urine protein in g/L
Time Frame: At Day 1 (pre-dose)
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
g/L | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)

52. Primary Outcome: Changes in Urinalysis Parameters
Description: Analysis was performed on urine samples collected at day 1 (post-dose) for the following parameter: urine protein in g/L. The change was calculated as difference between the day 1 (pre-dose) results and the day 1 (post-dose) results.
Time Frame: At Day 1 (post-dose)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of g/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of g/L | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

53. Primary Outcome: Changes in Urinalysis Parameters
Description: Analysis was performed on urine samples collected at day 8 (post-dose) for the following parameter: urine protein in g/L. The change was calculated as difference between the day 1 (pre-dose) results and the day 8 (post-dose) results.
Time Frame: At Day 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of g/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of g/L | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.047 (0.188) | 0.000 (0.000)

54. Primary Outcome: Changes in Urinalysis Parameters
Description: Analysis was performed on urine samples collected at day 29 (post-dose) for the following parameter: urine protein in g/L. The change was calculated as difference between the day 1 (pre-dose) results and the day 29 (post-dose) results.
Time Frame: At Day 29
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Difference of g/L
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Difference of g/L | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)

55. Primary Outcome: Number of Subjects With Abnormal Laboratory Parameter Values
Description: The abnormal laboratory parameters values were classified by the investigator as Normal (a value either low or high at baseline and normal post-baseline), High (a value either normal or low at baseline and high post-baseline), Low (a value either normal or high at baseline and low post-baseline) and No change.
Time Frame: At Day 1 (post-dose)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  ALT: Normal | 1 | 0 | 0 | 0 | 0
  ALT: High | 0 | 0 | 0 | 1 | 0
  ALT: Low | 0 | 0 | 0 | 0 | 0
  ALT: No change | 15 | 16 | 16 | 15 | 16
  AST: Normal | 0 | 0 | 0 | 0 | 0
  AST: High | 0 | 0 | 0 | 0 | 0
  AST: Low | 0 | 0 | 0 | 0 | 0
  AST: No change | 16 | 16 | 16 | 16 | 16
  Bicarbonate: Normal | 0 | 0 | 1 | 0 | 0
  Bicarbonate: High | 0 | 0 | 0 | 0 | 0
  Bicarbonate: Low | 0 | 0 | 0 | 0 | 0
  Bicarbonate: No change | 16 | 16 | 15 | 16 | 16
  BUN: Normal | 0 | 2 | 1 | 0 | 1
  BUN: High | 0 | 0 | 0 | 0 | 0
  BUN: Low | 1 | 0 | 0 | 3 | 0
  BUN: No change | 15 | 14 | 15 | 13 | 15
  CRP: Normal | 0 | 0 | 0 | 1 | 0
  CRP: High | 0 | 2 | 1 | 1 | 0
  CRP: Low | 0 | 0 | 0 | 0 | 0
  CRP: No change | 16 | 14 | 15 | 14 | 16
  Cl: Normal | 0 | 1 | 1 | 0 | 1
  Cl: High | 0 | 0 | 0 | 0 | 0
  Cl: Low | 0 | 0 | 0 | 1 | 1
  Cl: No change | 16 | 15 | 15 | 15 | 14
  CREA: Normal | 0 | 0 | 1 | 0 | 0
  CREA: High | 0 | 0 | 1 | 0 | 0
  CREA: Low | 0 | 0 | 0 | 0 | 0
  CREA: No change | 16 | 16 | 14 | 16 | 16
  K: Normal | 0 | 0 | 1 | 0 | 0
  K: High | 0 | 0 | 0 | 0 | 1
  K: Low | 0 | 0 | 0 | 0 | 0
  K: No change | 16 | 16 | 15 | 16 | 15
  Na: Normal | 0 | 4 | 0 | 0 | 1
  Na: High | 0 | 0 | 0 | 0 | 0
  Na: Low | 1 | 1 | 3 | 1 | 2
  Na: No change | 15 | 11 | 13 | 15 | 13
  Basophils: Normal | 1 | 0 | 0 | 0 | 0
  Basophils: High | 0 | 0 | 0 | 0 | 0
  Basophils: Low | 0 | 0 | 0 | 0 | 0
  Basophils: No change | 15 | 16 | 16 | 16 | 16
  Eosinophils: Normal | 0 | 1 | 0 | 0 | 0
  Eosinophils: High | 0 | 0 | 1 | 0 | 1
  Eosinophils: Low | 0 | 1 | 0 | 1 | 0
  Eosinophils: No change | 16 | 14 | 15 | 15 | 15
  RBC: Normal | 0 | 1 | 1 | 0 | 0
  RBC: High | 0 | 0 | 0 | 0 | 0
  RBC: Low | 0 | 0 | 0 | 0 | 0
  RBC: No change | 16 | 15 | 15 | 16 | 16
  Hematocrit: Normal | 0 | 0 | 0 | 0 | 0
  Hematocrit: High | 0 | 0 | 1 | 0 | 1
  Hematocrit: Low | 0 | 0 | 0 | 0 | 0
  Hematocrit: No change | 16 | 16 | 15 | 16 | 15
  Hemoglobin: Normal | 0 | 0 | 0 | 0 | 0
  Hemoglobin: High | 0 | 0 | 0 | 0 | 1
  Hemoglobin: Low | 0 | 0 | 0 | 0 | 0
  Hemoglobin: No change | 16 | 16 | 16 | 16 | 15
  Leukocytes: Normal | 1 | 0 | 0 | 0 | 0
  Leukocytes: High | 1 | 1 | 0 | 0 | 0
  Leukocytes: Low | 0 | 0 | 0 | 0 | 0
  Leukocytes: No change | 14 | 15 | 16 | 16 | 16
  Lymphocytes: Normal | 1 | 0 | 1 | 0 | 1
  Lymphocytes: High | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Low | 0 | 1 | 1 | 1 | 0
  Lymphocytes: No change | 15 | 15 | 14 | 15 | 15
  Monocytes: Normal | 2 | 4 | 1 | 2 | 1
  Monocytes: High | 0 | 0 | 0 | 0 | 0
  Monocytes: Low | 0 | 1 | 0 | 1 | 0
  Monocytes: No change | 14 | 11 | 15 | 13 | 15
  Neutrophils: Normal | 1 | 0 | 0 | 0 | 0
  Neutrophils: High | 2 | 1 | 0 | 0 | 0
  Neutrophils: Low | 0 | 0 | 0 | 0 | 0
  Neutrophils: No change | 13 | 15 | 16 | 16 | 16
  Platelets: Normal | 0 | 0 | 1 | 0 | 0
  Platelets: High | 0 | 0 | 0 | 0 | 0
  Platelets: Low | 0 | 2 | 0 | 1 | 0
  Platelets: No change | 16 | 14 | 15 | 15 | 16
  Urine RBC: Normal | 1 | 0 | 3 | 3 | 1
  Urine RBC: High | 0 | 1 | 0 | 1 | 0
  Urine RBC: Low | 0 | 0 | 0 | 0 | 0
  Urine RBC: No change | 15 | 15 | 13 | 12 | 15
  Urine Glucose: Normal | 0 | 0 | 0 | 0 | 0
  Urine Glucose: High | 0 | 0 | 0 | 0 | 0
  Urine Glucose: Low | 0 | 0 | 0 | 0 | 0
  Urine Glucose: No change | 16 | 16 | 16 | 16 | 16
  Urine Protein: Normal | 0 | 0 | 0 | 0 | 0
  Urine Protein: High | 0 | 0 | 0 | 0 | 0
  Urine Protein: Low | 0 | 0 | 0 | 0 | 0
  Urine Protein: No change | 16 | 16 | 16 | 16 | 16

56. Primary Outcome: Number of Subjects With Abnormal Laboratory Parameter Values
Description: as for outcome 55
Time Frame: At Day 8
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  ALT: Normal | 1 | 0 | 0 | 0 | 1
  ALT: High | 0 | 0 | 0 | 2 | 0
  ALT: Low | 0 | 0 | 0 | 0 | 0
  ALT: No change | 15 | 16 | 16 | 14 | 15
  AST: Normal | 0 | 0 | 0 | 0 | 0
  AST: High | 0 | 1 | 0 | 0 | 0
  AST: Low | 0 | 0 | 0 | 0 | 0
  AST: No change | 16 | 15 | 16 | 16 | 16
  Bicarbonate: Normal | 0 | 0 | 0 | 0 | 0
  Bicarbonate: High | 0 | 0 | 0 | 0 | 0
  Bicarbonate: Low | 0 | 0 | 0 | 0 | 0
  Bicarbonate: No change | 16 | 16 | 16 | 16 | 16
  BUN: Normal | 0 | 1 | 1 | 0 | 1
  BUN: High | 0 | 0 | 0 | 1 | 0
  BUN: Low | 1 | 0 | 0 | 1 | 1
  BUN: No change | 15 | 15 | 15 | 14 | 14
  CRP: Normal | 1 | 0 | 0 | 2 | 1
  CRP: High | 0 | 1 | 0 | 2 | 0
  CRP: Low | 0 | 0 | 0 | 0 | 0
  CRP: No change | 15 | 15 | 16 | 12 | 15
  Cl: Normal | 0 | 1 | 1 | 0 | 1
  Cl: High | 0 | 0 | 0 | 1 | 0
  Cl: Low | 1 | 0 | 0 | 4 | 2
  Cl: No change | 15 | 15 | 15 | 11 | 13
  CREA: Normal | 0 | 0 | 0 | 0 | 0
  CREA: High | 1 | 0 | 1 | 0 | 1
  CREA: Low | 0 | 0 | 0 | 0 | 0
  CREA: No change | 15 | 16 | 15 | 16 | 15
  K: Normal | 0 | 0 | 1 | 0 | 0
  K: High | 0 | 0 | 0 | 0 | 0
  K: Low | 0 | 0 | 0 | 0 | 0
  K: No change | 16 | 16 | 15 | 16 | 16
  Na: Normal | 0 | 3 | 4 | 1 | 0
  Na: High | 0 | 0 | 0 | 0 | 0
  Na: Low | 3 | 3 | 3 | 3 | 3
  Na: No change | 13 | 10 | 9 | 12 | 13
  Basophils: Normal | 1 | 0 | 0 | 0 | 0
  Basophils: High | 0 | 0 | 0 | 0 | 0
  Basophils: Low | 0 | 0 | 0 | 0 | 0
  Basophils: No change | 15 | 16 | 16 | 16 | 16
  Eosinophils: Normal | 0 | 1 | 0 | 0 | 0
  Eosinophils: High | 0 | 0 | 0 | 0 | 1
  Eosinophils: Low | 0 | 0 | 0 | 0 | 0
  Eosinophils: No change | 16 | 15 | 16 | 16 | 15
  RBC: Normal | 0 | 1 | 1 | 0 | 0
  RBC: High | 0 | 0 | 0 | 0 | 0
  RBC: Low | 0 | 0 | 1 | 0 | 0
  RBC: No change | 16 | 15 | 14 | 16 | 16
  Hematocrit: Normal | 0 | 0 | 0 | 0 | 0
  Hematocrit: High | 0 | 0 | 0 | 0 | 1
  Hematocrit: Low | 0 | 0 | 0 | 0 | 0
  Hematocrit: No change | 16 | 16 | 16 | 16 | 15
  Hemoglobin: Normal | 0 | 0 | 0 | 1 | 0
  Hemoglobin: High | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Low | 0 | 0 | 1 | 0 | 0
  Hemoglobin: No change | 16 | 16 | 15 | 15 | 16
  Leukocytes: Normal | 1 | 0 | 1 | 0 | 0
  Leukocytes: High | 1 | 0 | 0 | 0 | 0
  Leukocytes: Low | 0 | 1 | 1 | 0 | 0
  Leukocytes: No change | 14 | 15 | 14 | 16 | 16
  Lymphocytes: Normal | 1 | 1 | 1 | 0 | 2
  Lymphocytes: High | 0 | 0 | 1 | 0 | 0
  Lymphocytes: Low | 0 | 0 | 1 | 0 | 1
  Lymphocytes: No change | 15 | 15 | 13 | 16 | 13
  Monocytes: Normal | 1 | 3 | 0 | 1 | 1
  Monocytes: High | 0 | 0 | 0 | 0 | 0
  Monocytes: Low | 1 | 1 | 1 | 0 | 1
  Monocytes: No change | 14 | 12 | 15 | 15 | 14
  Neutrophils: Normal | 0 | 0 | 1 | 0 | 0
  Neutrophils: High | 1 | 0 | 0 | 0 | 0
  Neutrophils: Low | 0 | 1 | 0 | 0 | 0
  Neutrophils: No change | 15 | 15 | 15 | 16 | 16
  Platelets: Normal | 0 | 1 | 1 | 2 | 0
  Platelets: High | 0 | 0 | 0 | 0 | 0
  Platelets: Low | 0 | 0 | 0 | 0 | 0
  Platelets: No change | 16 | 15 | 15 | 14 | 16
  Urine RBC: Normal | 1 | 1 | 4 | 3 | 0
  Urine RBC: High | 0 | 2 | 0 | 1 | 0
  Urine RBC: Low | 0 | 0 | 0 | 0 | 0
  Urine RBC: No change | 15 | 13 | 12 | 12 | 16
  Urine Glucose: Normal | 0 | 0 | 0 | 0 | 0
  Urine Glucose: High | 0 | 0 | 0 | 0 | 0
  Urine Glucose: Low | 0 | 0 | 0 | 0 | 0
  Urine Glucose: No change | 16 | 16 | 16 | 16 | 16
  Urine Protein: Normal | 0 | 0 | 0 | 0 | 0
  Urine Protein: High | 0 | 0 | 0 | 1 | 0
  Urine Protein: Low | 0 | 0 | 0 | 0 | 0
  Urine Protein: No change | 16 | 16 | 16 | 15 | 16

57. Primary Outcome: Number of Subjects With Abnormal Laboratory Parameter Values
Description: as for outcome 55
Time Frame: At Day 29
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  ALT: Normal | 1 | 0 | 0 | 0 | 1
  ALT: High | 0 | 0 | 2 | 1 | 1
  ALT: Low | 0 | 0 | 0 | 0 | 0
  ALT: No change | 15 | 16 | 14 | 15 | 14
  AST: Normal | 0 | 0 | 0 | 0 | 0
  AST: High | 0 | 1 | 2 | 0 | 1
  AST: Low | 0 | 0 | 0 | 0 | 0
  AST: No change | 16 | 15 | 14 | 16 | 15
  Bicarbonate: Normal | 0 | 0 | 1 | 0 | 0
  Bicarbonate: High | 0 | 2 | 2 | 0 | 0
  Bicarbonate: Low | 0 | 0 | 0 | 0 | 0
  Bicarbonate: No change | 16 | 14 | 13 | 16 | 16
  BUN: Normal | 0 | 2 | 1 | 0 | 1
  BUN: High | 1 | 0 | 1 | 0 | 0
  BUN: Low | 0 | 0 | 0 | 1 | 2
  BUN: No change | 15 | 14 | 14 | 15 | 13
  CRP: Normal | 1 | 0 | 0 | 2 | 1
  CRP: High | 0 | 0 | 0 | 2 | 0
  CRP: Low | 0 | 0 | 0 | 0 | 0
  CRP: No change | 15 | 16 | 16 | 12 | 15
  Cl: Normal | 0 | 1 | 0 | 0 | 1
  Cl: High | 0 | 0 | 0 | 0 | 0
  Cl: Low | 1 | 1 | 1 | 2 | 2
  Cl: No change | 15 | 14 | 15 | 14 | 13
  CREA: Normal | 0 | 0 | 0 | 0 | 0
  CREA: High | 0 | 0 | 1 | 0 | 0
  CREA: Low | 0 | 0 | 0 | 0 | 0
  CREA: No change | 16 | 16 | 15 | 16 | 16
  K: Normal | 0 | 0 | 1 | 0 | 0
  K: High | 0 | 1 | 0 | 0 | 0
  K: Low | 0 | 0 | 0 | 0 | 0
  K: No change | 16 | 15 | 15 | 16 | 16
  Na: Normal | 0 | 5 | 5 | 0 | 2
  Na: High | 0 | 0 | 0 | 0 | 0
  Na: Low | 2 | 2 | 0 | 2 | 2
  Na: No change | 14 | 9 | 11 | 14 | 12
  Basophils: Normal | 1 | 0 | 0 | 0 | 0
  Basophils: High | 0 | 1 | 0 | 1 | 0
  Basophils: Low | 0 | 0 | 0 | 0 | 0
  Basophils: No change | 15 | 15 | 16 | 15 | 16
  Eosinophils: Normal | 0 | 1 | 0 | 0 | 0
  Eosinophils: High | 0 | 0 | 1 | 0 | 2
  Eosinophils: Low | 0 | 1 | 0 | 1 | 0
  Eosinophils: No change | 16 | 14 | 15 | 15 | 14
  RBC: Normal | 0 | 2 | 2 | 0 | 0
  RBC: High | 0 | 0 | 1 | 0 | 0
  RBC: Low | 0 | 0 | 0 | 0 | 0
  RBC: No change | 16 | 14 | 13 | 16 | 16
  Hematocrit: Normal | 0 | 0 | 0 | 0 | 0
  Hematocrit: High | 1 | 2 | 0 | 0 | 0
  Hematocrit: Low | 0 | 0 | 0 | 0 | 0
  Hematocrit: No change | 15 | 14 | 16 | 16 | 16
  Hemoglobin: Normal | 0 | 0 | 0 | 1 | 0
  Hemoglobin: High | 1 | 0 | 1 | 0 | 0
  Hemoglobin: Low | 0 | 0 | 0 | 0 | 0
  Hemoglobin: No change | 15 | 16 | 15 | 15 | 16
  Leukocytes: Normal | 1 | 0 | 1 | 0 | 0
  Leukocytes: High | 1 | 0 | 0 | 0 | 0
  Leukocytes: Low | 0 | 0 | 0 | 0 | 0
  Leukocytes: No change | 14 | 16 | 15 | 16 | 16
  Lymphocytes: Normal | 1 | 1 | 1 | 0 | 2
  Lymphocytes: High | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Low | 1 | 0 | 0 | 0 | 0
  Lymphocytes: No change | 14 | 15 | 15 | 16 | 14
  Monocytes: Normal | 2 | 3 | 0 | 0 | 0
  Monocytes: High | 0 | 0 | 0 | 0 | 0
  Monocytes: Low | 0 | 0 | 0 | 0 | 0
  Monocytes: No change | 14 | 13 | 16 | 16 | 16
  Neutrophils: Normal | 1 | 0 | 1 | 0 | 0
  Neutrophils: High | 1 | 0 | 0 | 1 | 0
  Neutrophils: Low | 0 | 0 | 0 | 0 | 0
  Neutrophils: No change | 14 | 16 | 15 | 15 | 16
  Platelets: Normal | 0 | 1 | 1 | 2 | 0
  Platelets: High | 1 | 0 | 0 | 0 | 0
  Platelets: Low | 0 | 0 | 1 | 1 | 0
  Platelets: No change | 15 | 15 | 14 | 13 | 16
  Urine RBC: Normal | 2 | 1 | 4 | 4 | 2
  Urine RBC: High | 0 | 3 | 2 | 2 | 0
  Urine RBC: Low | 0 | 0 | 0 | 0 | 0
  Urine RBC: No change | 14 | 12 | 10 | 10 | 14
  Urine Glucose: Normal | 0 | 0 | 0 | 0 | 0
  Urine Glucose: High | 0 | 0 | 0 | 0 | 0
  Urine Glucose: Low | 0 | 0 | 0 | 0 | 0
  Urine Glucose: No change | 16 | 16 | 16 | 16 | 16
  Urine Protein: Normal | 0 | 0 | 0 | 0 | 0
  Urine Protein: High | 0 | 0 | 0 | 0 | 0
  Urine Protein: Low | 0 | 0 | 0 | 0 | 0
  Urine Protein: No change | 16 | 16 | 16 | 16 | 16

58. Primary Outcome: Number of Subjects With Abnormal Laboratory Parameter Values
Description: The abnormal laboratory parameters values were defined following the FDA CBER Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" dated September 2007, or the institution's normal ranges if they differ from CBER guidance
Time Frame: At Day 1 (post-dose)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  ALT: None | 16 | 16 | 16 | 15 | 15
  ALT: Grade 1 | 0 | 0 | 0 | 1 | 1
  ALT: Grade 2 | 0 | 0 | 0 | 0 | 0
  ALT: Grade 3 | 0 | 0 | 0 | 0 | 0
  ALT: Grade 4 | 0 | 0 | 0 | 0 | 0
  AST: None | 16 | 16 | 16 | 16 | 16
  AST: Grade 1 | 0 | 0 | 0 | 0 | 0
  AST: Grade 2 | 0 | 0 | 0 | 0 | 0
  AST: Grade 3 | 0 | 0 | 0 | 0 | 0
  AST: Grade 4 | 0 | 0 | 0 | 0 | 0
  BUN: None | 16 | 16 | 16 | 16 | 16
  BUN: Grade 1 | 0 | 0 | 0 | 0 | 0
  BUN: Grade 2 | 0 | 0 | 0 | 0 | 0
  BUN: Grade 3 | 0 | 0 | 0 | 0 | 0
  BUN: Grade 4 | 0 | 0 | 0 | 0 | 0
  CREA: None | 16 | 16 | 16 | 16 | 16
  CREA: Grade 1 | 0 | 0 | 0 | 0 | 0
  CREA: Grade 2 | 0 | 0 | 0 | 0 | 0
  CREA: Grade 3 | 0 | 0 | 0 | 0 | 0
  CREA: Grade 4 | 0 | 0 | 0 | 0 | 0
  HGB: None | 12 | 13 | 12 | 8 | 13
  HGB: Grade 1 | 4 | 3 | 4 | 8 | 3
  HGB: Grade 2 | 0 | 0 | 0 | 0 | 0
  HGB: Grade 3 | 0 | 0 | 0 | 0 | 0
  HGB: Grade 4 | 0 | 0 | 0 | 0 | 0
  Leukocytes: None | 16 | 16 | 16 | 16 | 16
  Leukocytes: Grade 1 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 2 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 3 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelets: None | 15 | 15 | 16 | 15 | 15
  Platelets: Grade 1 | 0 | 1 | 0 | 1 | 1
  Platelets: Grade 2 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 3 | 1 | 0 | 0 | 0 | 0
  Platelets: Grade 4 | 0 | 0 | 0 | 0 | 0

59. Primary Outcome: Number of Subjects With Abnormal Laboratory Parameter Values
Description: as for outcome 58
Time Frame: At Day 8
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  ALT: None | 16 | 16 | 16 | 15 | 16
  ALT: Grade 1 | 0 | 0 | 0 | 1 | 0
  ALT: Grade 2 | 0 | 0 | 0 | 0 | 0
  ALT: Grade 3 | 0 | 0 | 0 | 0 | 0
  ALT: Grade 4 | 0 | 0 | 0 | 0 | 0
  AST: None | 16 | 15 | 16 | 16 | 16
  AST: Grade 1 | 0 | 1 | 0 | 0 | 0
  AST: Grade 2 | 0 | 0 | 0 | 0 | 0
  AST: Grade 3 | 0 | 0 | 0 | 0 | 0
  AST: Grade 4 | 0 | 0 | 0 | 0 | 0
  BUN: None | 16 | 16 | 16 | 16 | 16
  BUN: Grade 1 | 0 | 0 | 0 | 0 | 0
  BUN: Grade 2 | 0 | 0 | 0 | 0 | 0
  BUN: Grade 3 | 0 | 0 | 0 | 0 | 0
  BUN: Grade 4 | 0 | 0 | 0 | 0 | 0
  CREA: None | 16 | 16 | 16 | 16 | 16
  CREA: Grade 1 | 0 | 0 | 0 | 0 | 0
  CREA: Grade 2 | 0 | 0 | 0 | 0 | 0
  CREA: Grade 3 | 0 | 0 | 0 | 0 | 0
  CREA: Grade 4 | 0 | 0 | 0 | 0 | 0
  HGB: None | 9 | 12 | 8 | 12 | 13
  HGB: Grade 1 | 7 | 4 | 7 | 4 | 3
  HGB: Grade 2 | 0 | 0 | 1 | 0 | 0
  HGB: Grade 3 | 0 | 0 | 0 | 0 | 0
  HGB: Grade 4 | 0 | 0 | 0 | 0 | 0
  Leukocytes: None | 15 | 15 | 15 | 16 | 16
  Leukocytes: Grade 1 | 1 | 1 | 1 | 0 | 0
  Leukocytes: Grade 2 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 3 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelets: None | 15 | 16 | 16 | 16 | 16
  Platelets: Grade 1 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 2 | 1 | 0 | 0 | 0 | 0
  Platelets: Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 4 | 0 | 0 | 0 | 0 | 0

60. Primary Outcome: Number of Subjects With Abnormal Laboratory Parameter Values
Description: as for outcome 58
Time Frame: At Day 29
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Participants
  ALT: None | 16 | 16 | 14 | 15 | 16
  ALT: Grade 1 | 0 | 0 | 2 | 1 | 0
  ALT: Grade 2 | 0 | 0 | 0 | 0 | 0
  ALT: Grade 3 | 0 | 0 | 0 | 0 | 0
  ALT: Grade 4 | 0 | 0 | 0 | 0 | 0
  AST: None | 16 | 15 | 14 | 16 | 15
  AST: Grade 1 | 0 | 1 | 2 | 0 | 1
  AST: Grade 2 | 0 | 0 | 0 | 0 | 0
  AST: Grade 3 | 0 | 0 | 0 | 0 | 0
  AST: Grade 4 | 0 | 0 | 0 | 0 | 0
  BUN: None | 16 | 16 | 15 | 16 | 16
  BUN: Grade 1 | 0 | 0 | 1 | 0 | 0
  BUN: Grade 2 | 0 | 0 | 0 | 0 | 0
  BUN: Grade 3 | 0 | 0 | 0 | 0 | 0
  BUN: Grade 4 | 0 | 0 | 0 | 0 | 0
  CREA: None | 16 | 16 | 16 | 16 | 16
  CREA: Grade 1 | 0 | 0 | 0 | 0 | 0
  CREA: Grade 2 | 0 | 0 | 0 | 0 | 0
  CREA: Grade 3 | 0 | 0 | 0 | 0 | 0
  CREA: Grade 4 | 0 | 0 | 0 | 0 | 0
  HGB: None | 10 | 14 | 13 | 11 | 10
  HGB: Grade 1 | 6 | 2 | 3 | 5 | 6
  HGB: Grade 2 | 0 | 0 | 0 | 0 | 0
  HGB: Grade 3 | 0 | 0 | 0 | 0 | 0
  HGB: Grade 4 | 0 | 0 | 0 | 0 | 0
  Leukocytes: None | 16 | 16 | 16 | 16 | 16
  Leukocytes: Grade 1 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 2 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 3 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Grade 4 | 0 | 0 | 0 | 0 | 0
  Platelets: None | 15 | 16 | 16 | 16 | 16
  Platelets: Grade 1 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 2 | 1 | 0 | 0 | 0 | 0
  Platelets: Grade 3 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 4 | 0 | 0 | 0 | 0 | 0

61. Primary Outcome: Human Complement Serum Bactericidal Assay (hSBA) Geometric Mean Titers (GMTs) Against N. Meningitidis Serogroup C (MenC)
Description: The antibody concentrations were assessed by hSBA directed against MenC serogroup and expressed as GMTs.
Time Frame: At Day 1 (pre-dose)
Population: Analysis was performed on the Per Protocol Set (PPS) which included subjects who received a study vaccination and provided efficacy or immunogenicity data at relevant time points and who were not excluded due to reasons defined prior to unbliding or analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Titer | 11.40 [6.23 to 20.86] | 8.52 [4.66 to 15.59] | 6.09 [3.33 to 11.13] | 5.23 [2.86 to 9.57] | 6.17 [3.37 to 11.28]

62. Primary Outcome: hSBA GMTs Against N. Meningitidis Serogroup C (MenC)
Description: The antibody concentrations were assessed by hSBA directed against MenC serogroup and expressed as GMTs.
Time Frame: At Day 29
Population: Analysis was performed on the PPS which included subjects who received a study vaccination and provided efficacy or immunogenicity data at relevant time points and who were not excluded due to reasons defined prior to unbliding or analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Titer | 96.61 [34.97 to 266.89] | 55.05 [20.19 to 150.06] | 101.77 [37.34 to 277.39] | 56.31 [20.55 to 154.29] | 70.38 [25.83 to 191.79]

63. Primary Outcome: Geometric Mean Ratio (GMR) of the Titers of Antibodies Measured by hSBA Against MenC Serogroup
Description: GMR of GMTs of antibodies against MenC was evaluated at Day 29 relative to Day 1 (pre-dose).
Time Frame: At Day 29
Population: Analysis was performed on the PPS which included subjects who received a study vaccination and provided efficacy or immunogenicity data at relevant time points and who were not excluded due to reasons defined prior to unblinding or analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Ratio | 8.70 [2.77 to 27.36] | 6.52 [2.08 to 20.51] | 16.56 [5.27 to 52.07] | 10.57 [3.36 to 33.23] | 11.32 [3.60 to 35.57]

64. Secondary Outcome: hSBA GMTs Against N. Meningitidis Serogroup C (MenC)
Description: The antibody concentrations were assessed by hSBA directed against MenC and expressed as GMTs.
Time Frame: At Day 8 and Day 181
Population: as for outcome 63
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Titer
  Day 8 | 30.86 [12.61 to 75.50] | 12.18 [5.04 to 29.47] | 13.58 [5.61 to 32.87] | 15.47 [6.20 to 38.65] | 21.30 [8.80 to 51.53]
  Day 181: number analyzed (Participants) | 16 | 16 | 16 | 16 | 15
  Day 181 | 98.79 [49.66 to 196.52] | 68.89 [34.94 to 135.83] | 83.59 [42.40 to 164.78] | 63.13 [31.91 to 124.91] | 59.67 [29.61 to 120.27]

65. Secondary Outcome: GMR of the GMTs of Antibodies Measured by hSBA Against MenC Serogroup
Description: GMR of GMTs of antibodies against MenC serogroup was evaluated at Day 8 and Day 181 relative to Day 1 (pre-dose).
Time Frame: At Day 8 and Day 181
Population: as for outcome 63
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Ratio
  Day 8/Day 1 | 2.93 [1.07 to 8.03] | 1.47 [0.54 to 4.02] | 2.16 [0.79 to 5.91] | 2.64 [0.93 to 7.48] | 3.35 [1.22 to 9.17]
  Day 181/Day 1: number analyzed (Participants) | 16 | 16 | 16 | 16 | 15
  Day 181/Day 1 | 9.29 [3.98 to 21.69] | 8.30 [3.55 to 19.37] | 13.40 [5.74 to 31.28] | 11.51 [4.93 to 26.87] | 9.53 [3.97 to 22.87]

66. Secondary Outcome: Percentage of Subjects With hSBA Seroresponse Against N. Meningitidis Serogroup C (MenC).
Description: The percentage of subjects who achieved hSBA seroresponse against MenC serogroup was evaluated at Day 8, Day 29 and Day 181 after vaccination. Seroresponse was defined as a post vaccination hSBA ≥ 8 for subjects with a baseline hSBA lower than (<) 4 or had an increase of at least 4 times the baseline hSBA level for subjects with pre vaccination hSBA ≥ 4.
Time Frame: At Day 8, Day 29 and Day 181
Population: as for outcome 63
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Percentage of subjects
  Day 8: number analyzed (Participants) | 16 | 16 | 16 | 15 | 16
  Day 8 | 31.3 [11.0 to 58.7] | 37.5 [15.2 to 64.6] | 31.3 [11.0 to 58.7] | 33.3 [11.8 to 61.6] | 37.5 [15.2 to 64.6]
  Day 29 | 75.0 [47.6 to 92.7] | 56.3 [29.9 to 80.2] | 81.3 [54.4 to 96.0] | 68.8 [41.3 to 89.0] | 75.0 [47.6 to 92.7]
  Day 181: number analyzed (Participants) | 16 | 16 | 16 | 16 | 15
  Day 181 | 75.0 [47.6 to 92.7] | 56.3 [29.9 to 80.2] | 87.5 [61.7 to 98.4] | 75.0 [47.6 to 92.7] | 80.0 [51.9 to 95.7]

67. Secondary Outcome: Concentrations of Antibodies Against MenC Serogroup Measured by Enzyme Linked Immunosorbent Assay (ELISA)
Description: The antibody concentrations were assessed by ELISA and expressed as Geometric Mean Concentrations (GMCs) in microgram per mililiter (μg/mL).
Time Frame: At Day 1 (pre-dose), Day 8, Day 29 and Day 181
Population: as for outcome 63
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
μg/mL
  Day 1 (pre-dose) | 0.287 [0.124 to 0.664] | 0.407 [0.176 to 0.942] | 0.207 [0.089 to 0.479] | 0.107 [0.046 to 0.249] | 0.199 [0.086 to 0.462]
  Day 8 | 2.005 [0.980 to 4.101] | 2.169 [1.052 to 4.472] | 1.668 [0.817 to 3.406] | 2.897 [1.400 to 5.997] | 1.445 [0.708 to 2.951]
  Day 29 | 15.946 [9.265 to 27.444] | 12.753 [7.364 to 22.086] | 19.322 [11.242 to 33.210] | 21.944 [12.636 to 38.107] | 9.207 [5.356 to 15.827]
  Day 181: number analyzed (Participants) | 16 | 16 | 16 | 16 | 15
  Day 181 | 5.201 [3.218 to 8.406] | 5.556 [3.419 to 9.027] | 7.131 [4.416 to 11.513] | 7.570 [4.644 to 12.339] | 3.432 [2.093 to 5.628]

68. Secondary Outcome: Percentage of Subjects With at Least a 4-fold Increase in Antibody Concentrations to MenC as Measured by ELISA
Description: The percentage of subjects with at least a 4-fold increase in antibody concentrations to MenC serogroup as measured by ELISA were analysed at day 8, 29 and 181 relative to Day 1 (pre-dose).
Time Frame: At Day 8, Day 29 and Day 181
Population: as for outcome 63
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
Percentage of subjects
  Day 8 | 68.8 [41.3 to 89.0] | 50.0 [24.7 to 75.3] | 68.8 [41.3 to 89.0] | 68.8 [41.3 to 89.0] | 62.5 [35.4 to 84.8]
  Day 29 | 93.8 [69.8 to 99.8] | 81.3 [54.4 to 96.0] | 100.0 [79.4 to 100.0] | 100.0 [79.4 to 100.0] | 87.5 [61.7 to 98.4]
  Day 181: number analyzed (Participants) | 16 | 16 | 16 | 16 | 15
  Day 181 | 87.5 [61.7 to 98.4] | 75.0 [47.6 to 92.7] | 100.0 [79.4 to 100.0] | 100.0 [79.4 to 100.0] | 86.7 [59.5 to 98.3]

ADVERSE EVENTS:
Time Frame: Solicited local and systemic AEs were collected from Day 1 (30 minutes) until Day 14 after vaccination. Unsolicited AEs were collected from Day 1 to Day 29. Serious AEs were collected from day 1 to study completion date (Day 366).
Arm/Group | LHD153R Formulation 1 Group | LHD153R Formulation 2 Group | LHD153R Formulation 3 Group | LHD153R Formulation 4 Group | MenC Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 1/16
Other Adverse Events (participants affected / at risk) | 16/16 | 16/16 | 16/16 | 16/16 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LHD153R Formulation 1 Group (N=16) | LHD153R Formulation 2 Group (N=16) | LHD153R Formulation 3 Group (N=16) | LHD153R Formulation 4 Group (N=16) | MenC Group (N=16)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LHD153R Formulation 1 Group (N=16) | LHD153R Formulation 2 Group (N=16) | LHD153R Formulation 3 Group (N=16) | LHD153R Formulation 4 Group (N=16) | MenC Group (N=16)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 2 (2) | 1 (1) | 3 (4) | 3 (4)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Induration (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — This AE was recorded as a solicited local AE
Pain (General disorders) | 16 (214) | 16 (216) | 16 (213) | 16 (216) | 16 (210) — This AE was recorded as a solicited local AE
Swelling (General disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) — This AE was recorded as a solicited local AE
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — This AE was reported as an unsolicited AE
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — This AE was reported as an unsolicited AE
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (General disorders) | 1 (3) | 1 (2) | 0 (0) | 4 (6) | 0 (0) — This adverse event was recorded as a systemic adverse event
Chills (General disorders) | 0 (0) | 2 (4) | 1 (1) | 4 (9) | 1 (1) — This AE was recorded as a systemic adverse event
Diarrhea (General disorders) | 1 (2) | 0 (0) | 1 (2) | 3 (5) | 0 (0) — This AE was recorded as a systemic AE
Fatigue (General disorders) | 3 (10) | 2 (10) | 3 (3) | 6 (25) | 3 (3) — This AE was recorded as a systemic AE
Fever (General disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (11) | 0 (0) — This AE was recorded as a systemic AE
Headache (General disorders) | 6 (13) | 7 (21) | 5 (8) | 5 (18) | 10 (15) — This AE was recorded as a systemic AE
Loss of Appetite (General disorders) | 1 (2) | 1 (3) | 2 (2) | 4 (15) | 0 (0) — This AE was recorded as a systemic AE
Myalgia (General disorders) | 1 (3) | 1 (3) | 0 (0) | 5 (12) | 3 (3) — This AE was recorded as a systemic AE
Nausea (General disorders) | 1 (1) | 2 (4) | 2 (2) | 3 (7) | 1 (1) — This AE was recorded as a systemic AE
Rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — This AE was recorded as a systemic AE
Urticaria (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — This AE was recorded as a solicited AE
Vomiting (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) — This AE was reported as a systemic AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2014-06-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT02639351/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02639351/SAP_001.pdf